CLINICAL TRIAL: NCT04322201
Title: Continuous Passive Paracentesis Versus Large Volume Paracentesis in the Prevention and Treatment of Intra-abdominal Hypertension and Abdominal Compartment Syndrome in the Critically Ill Cirrhotic Patient With Ascites
Brief Title: Continuous Passive Paracentesis for Intra-abdominal Hypertension
Acronym: COPPTRIAHL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Hospitalar de Lisboa Central (Other)
Collaborators: NOVA Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHULC.CI.450.2019
Record Dates: First submitted 2019-12-20; First posted 2020-03-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Ascites Hepatic; Cirrhosis, Liver; Hypertension, Intraabdominal; Critical Illness; Paracentesis
Keywords: Hepatic Ascites; Liver Cirrhosis; Intraabdominal Hypertension; Paracentesis; Puncture and Drainage; Critical Illness; acute-on-chronic liver failure
MeSH Terms: conditions — Liver Cirrhosis; Intra-Abdominal Hypertension; Critical Illness; Acute-On-Chronic Liver Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group - Continuous passive paracentesis (Experimental): Ultrasound-guided placement of an intra-abdominal double lumen central venous catheter, using aseptic Seldinger technique, for continuous drainage of ascitic fluid up to 7 days in Intensive Care.
  Interventions: Device: continuous drainage of ascitic fluid using an intra-abdominal double lumen central venous catheter
- Control group - Large volume paracentesis (Active Comparator): Ultrasound-guided intermittent large-volume paracentesis through 14 Gauge catheter performed and repeated during ICU stay according to standard-of-care clinical practice.
  Interventions: Procedure: Ultrasound-guided intermittent large-volume paracentesis

INTERVENTIONS:
Device: continuous drainage of ascitic fluid using an intra-abdominal double lumen central venous catheter — Ultrasound-guided placement of an intra-abdominal double lumen central venous catheter, using aseptic Seldinger technique, for continuous drainage of ascitic fluid up to 7 days in Intensive Care
  Other Names: continuous passive paracentesis
  Arms: Intervention group - Continuous passive paracentesis
Procedure: Ultrasound-guided intermittent large-volume paracentesis — Ultrasound-guided intermittent large-volume paracentesis through 14 Gauge catheter
  Other Names: intermittent passive paracentesis
  Arms: Control group - Large volume paracentesis

SUMMARY:
Liver cirrhosis patients in Intensive Care present intra-abdominal hypertension and this is an independent risk factor for increased organ disfunction and mortality.

Patients will be randomized into intermittent or continuous passive paracentesis and the clinical results of these two strategies for preventing and treating intra-abdominal hypertension will compared.

DETAILED DESCRIPTION:
Intra-abdominal hypertension is an independent risk factors for increased mortality in Intensive Care patients and is highly prevalent in the critically ill cirrhotic patient. This study compares two strategies in minimizing intra-abdominal pressure and optimizing abdominal perfusion pressure in the prevention and treatment of intra-abdominal hypertension associated morbidity and mortality. Critically ill cirrhotic patients will be allocated into a standard-of-care large-volume paracentesis group (control) and a continuous passive paracentesis (intervention) group using randomization. Results will assess renal function and multi-organ function using standard clinical scales and vital outcomes.

ELIGIBILITY:
Inclusion Criteria:

* liver cirrhosis diagnosis with ascites
* ICU admission for medical reason

Exclusion Criteria:

* prior liver transplant
* haemorrhagic ascites
* extreme severity: CLIF-SOFA number of organ failures 5 or more
* less than 24 hours of ICU stay
* Any of the following conditions at 24 hours of ICU stay:

  i. Hemorrhagic shock with active uncontrolled bleeding ii. Refractory shock (MAP<60mmHg) with multiple vasopressors iii. Predictably short ICU stay (<72 hours) iv. Therapeutic futility determined by the medical staff

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-11-02 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Renal function - creatinine clearance | intensive care stay up to 7 days
  estimated and measured creatinine clearance (mL/min)
Renal function - urine output | intensive care stay up to 7 days
  measured urine output (mL/min)
Renal function - renal replacement therapy | intensive care stay up to 7 days
  number of renal replacement therapy days
Multi-organ disfunction | intensive care stay up to 7 days
  Clinical multi-organ disfunction as assessed by severity scores: Sequencial Organ Failure Assessement (SOFA) and Chronic Liver Failure-SOFA (CLIF-SOFA). Both scores range [0-24] and higher scores reflect more severe organ dysfunctions and worse outcomes.

SECONDARY OUTCOMES:
ICU Mortality rate | from admission into the ICU up to 30 days onwards
  Mortality rate until discharge from the ICU
in hospital Mortality rate | from admission into the ICU up to 60 days onwards
  Mortality rate until discharge from hospital admission
30 days Mortality rate | from admission into the ICU up to 30 days onwards
  Mortality rate up to 30 days from ICU admission
Emergent liver transplant rate | from admission into the ICU up to 28 days onwards
  liver transplant rate up to 28 days after ICU admission

OTHER OUTCOMES:
ICU length-of-stay | from admission into the ICU up to 28 days
  days in Intensive Care Unit
Hospital length-of-stay | from admission into the ICU up to 60 days onwards
  days of Hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Rui A Pereira, MD, MSc, Principal Investigator — Centro Hospitalar de Lisboa Central
Locations (1):
- UCIP7 - Centro Hospitalar Universitário de Lisboa Central, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caldwell J, Edriss H, Nugent K. Chronic peritoneal indwelling catheters for the management of malignant and nonmalignant ascites. Proc (Bayl Univ Med Cent). 2018 Jun 1;31(3):297-302. doi: 10.1080/08998280.2018.1461525. eCollection 2018 Jul. PMID 29904292
- [Background] Kyoung KH, Hong SK. The duration of intra-abdominal hypertension strongly predicts outcomes for the critically ill surgical patients: a prospective observational study. World J Emerg Surg. 2015 May 30;10:22. doi: 10.1186/s13017-015-0016-7. eCollection 2015. PMID 26056530
- [Background] Kirkpatrick AW, Roberts DJ, De Waele J, Jaeschke R, Malbrain ML, De Keulenaer B, Duchesne J, Bjorck M, Leppaniemi A, Ejike JC, Sugrue M, Cheatham M, Ivatury R, Ball CG, Reintam Blaser A, Regli A, Balogh ZJ, D'Amours S, Debergh D, Kaplan M, Kimball E, Olvera C; Pediatric Guidelines Sub-Committee for the World Society of the Abdominal Compartment Syndrome. Intra-abdominal hypertension and the abdominal compartment syndrome: updated consensus definitions and clinical practice guidelines from the World Society of the Abdominal Compartment Syndrome. Intensive Care Med. 2013 Jul;39(7):1190-206. doi: 10.1007/s00134-013-2906-z. Epub 2013 May 15. PMID 23673399
- [Result] Al-Dorzi HM, Tamim HM, Rishu AH, Aljumah A, Arabi YM. Intra-abdominal pressure and abdominal perfusion pressure in cirrhotic patients with septic shock. Ann Intensive Care. 2012 Jul 5;2 Suppl 1(Suppl 1):S4. doi: 10.1186/2110-5820-2-S1-S4. Epub 2012 Jul 5. PMID 22873420
- [Derived] Pereira RA, Virella D, Perdigoto R, Marcelino P, Saliba F, Germano N. Continuous passive paracentesis versus large-volume paracentesis in the prevention and treatment of intra-abdominal hypertension in the critically ill cirrhotic patient with ascites (COPPTRIAHL): study protocol for a randomized controlled trial. Trials. 2023 Aug 15;24(1):534. doi: 10.1186/s13063-023-07541-4. PMID 37582719